CLINICAL TRIAL: NCT02444793
Title: A PHASE 1B STUDY OF PF-05082566 IN COMBINATION WITH MOGAMULIZUMAB (KW-0761) IN PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study of PF-05082566 In Combination With Mogamulizumab In Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to marginal efficacy and change in sponsor prioritization. The combination had a manageable safety profile.
Sponsor: Pfizer (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B1641004
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Advanced/Metastatic Solid Tumors
MeSH Terms: interventions — utomilumab; mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-05082566 + KW-0761 (Experimental): During Parts 1 & 2 Mogamulizumab and PF-05082566 will be administered at appropriate intervals. Part 1: PF-05082566 dose escalation; increased doses of PF-05082566 IV are administered with mogamulizumab IV. Part 2: patients will be treated with the maximum tolerated dose established in Phase 1 for the combination.
  Interventions: Drug: PF-05082566; Drug: KW-0761

INTERVENTIONS:
Drug: PF-05082566 — Part 1: PF-05082566 dose escalation; Increased doses of PF-05082566 IV are administered at appropriate intervals. Part 2: MTD of PF-05082566 IV established in Part 1 is administered.
Drug: KW-0761 — Part 1: KW-0761 IV administered at appropriate intervals. Part 2: KW-0761 IV administered at appropriate intervals at the MTD dose for the combination.
  Other Names: KW-0761= Mogamulizumab or POTELIGEO®

SUMMARY:
This study is a Phase 1b, open label, multi center, multi-dose trial designed to estimate the maximum tolerated dose (MTD) and select the recommended dose for phase 2 (RP2D) investigations of PF- 05082566 in combination with KW-0761 (mogamulizumab) in patients with advanced solid tumors. Once the MTD of PF-05082566 administered in combination with KW-0761 is estimated (dose finding), one or more expansion cohorts of patients with selected advanced solid tumors (dose-expansion ) will be enrolled to further characterize the combination in term of safety profile, anti tumor activity, pharmacokinetics, pharmacodynamics and biomarkers modulation.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced/metastatic solid tumor malignancy. Dose Finding Cohorts: Tumor types will be limited to CRC, SCCHN, squamous NSCLC, bladder, or ovarian carcinomas which have progressed on standard therapy, or for which no standard therapy is available.
* Measurable disease by RECIST version 1.1.
* For Expansion Cohorts only: patients must have tumor accessible for biopsies (core needle biopsy or excision preferred).
* Age 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone marrow, renal and liver function.
* Serum/urine pregnancy test (for females of childbearing potential) negative at screening and before the patient will receive the study treatment.
* Male and female patients of childbearing potential and at risk for pregnancy must agree to use two (2) highly effective methods of contraception throughout the study and for 60 days after the last dose of assigned study treatment.

Exclusion Criteria:

* Active central nervous system primary or secondary malignancies, active seizure disorder, spinal cord compression, or carcinomatous meningitis.
* Therapeutic or experimental monoclonal antibodies in last 60 days prior registration.
* Systemic anticancer therapy or major surgery within 28 days prior to registration. In absence of toxicity from prior systemic anticancer therapy, 5 half-lives since completion of prior systemic anticancer therapy is allowed.
* Systemic steroids, any other form of immunosuppressive therapy or radiation therapy within 14 days prior to registration.
* Live vaccine within 30 days prior to registration.
* Severe hypersensitivity reaction to treatment with another monoclonal antibody, known or suspected hypersensitivity to study drugs or any component of their formulation.
* History of autoimmune disease or known inflammatory bowel disease.
* Uncontrolled hypertension (blood pressure >150/100 mmHg despite optimal medical therapy) or any of the following within 12 months prior to registration: myocardial infarction, congenital long QT syndrome, torsade de points, arrhythmias, right bundle branch block and left anterior hemiblock uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, ongoing NCICTCAE Grade 2 cardiac dysrhythmias, atrial fibrillation or QTcF interval >470 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Michael J Pishvaian, MD, PhD, Principal Investigator — Georgetown University; Esra E Cohen, MD, Principal Investigator — University of California, San Diego; Dale R Shepard, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (21):
- United States (21):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - La Jolla(Thornton Hospital), La Jolla, California
  - University Of California / San Diego Moores Cancer Center, La Jolla, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Henry Ford Hospital Research Pharmacy, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - UNC Cancer Hospital Infusion Pharmacy, Chapel Hill, North Carolina
  - UNC Hospitals, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Sanford Research, Sioux Falls, South Dakota
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Cohen EEW, Pishvaian MJ, Shepard DR, Wang D, Weiss J, Johnson ML, Chung CH, Chen Y, Huang B, Davis CB, Toffalorio F, Thall A, Powell SF. A phase Ib study of utomilumab (PF-05082566) in combination with mogamulizumab in patients with advanced solid tumors. J Immunother Cancer. 2019 Dec 4;7(1):342. doi: 10.1186/s40425-019-0815-6. PMID 31801624
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1641004&StudyName=A%20Phase%201b%20Study%20Of%20Pf-05082566%20In%20Combination%20With%20Mogamulizumab%20%28kw-0761%29%20In%20Patients%20With%20Advanced%20Solid%20Tumors
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1641004&StudyName=A+Phase+1b+Study+Of+Pf-05082566+In+Combination+With+Mogamulizumab+%28kw-0761%29+In+Patients+With+Advanced+Solid+Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion every 4 weeks on Day 1 of each cycle at 1.2 mg/kg. Mogamulizumab was administered as a 1-hour intravenous infusion weekly for 4 consecutive weeks (Days 1, 8, 15 and 22) followed by biweekly dosing (Days 1 and 15) at 1 mg/kg.
- PF-05082566 100 mg + Mogamulizumab 1 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion every 4 weeks on Day 1 of each cycle at 100 mg. Mogamulizumab was administered as a 1-hour intravenous infusion weekly for 4 consecutive weeks (Days 1, 8, 15 and 22) followed by biweekly dosing (Days 1 and 15) at 1 mg/kg.
- PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion every 4 weeks on Day 1 of each cycle at 2.4 mg/kg. Mogamulizumab was administered as a 1-hour intravenous infusion weekly for 4 consecutive weeks (Days 1, 8, 15 and 22) followed by biweekly dosing (Days 1 and 15) at 1 mg/kg.
- PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg: PF-05082566 was administered as a 1-hour intravenous infusion every 4 weeks on Day 1 of each cycle at 5 mg/kg. Mogamulizumab was administered as a 1-hour intravenous infusion weekly for 4 consecutive weeks (Days 1, 8, 15 and 22) followed by biweekly dosing (Days 1 and 15) at 1 mg/kg.
Period: Overall Study
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Started | 11 | 6 | 4 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 11 | 6 | 4 | 3
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0
Not completed — Death | 0 | 3 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0
Not completed — Objective progression or relapse | 9 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Included all enrolled participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg | Total
Number analyzed (Participants) | 11 | 6 | 4 | 3 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (4.9) | 66.2 (8.6) | 67.8 (4.0) | 62.7 (8.7) | 63.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 5
  Male | 10 | 5 | 2 | 2 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 6 | 3 | 1 | 19
  Black | 2 | 0 | 1 | 1 | 4
  Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: DLTs was defined as any of the following adverse events (AEs) according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 at first 2 Cycles. Hematologic: (1) Grade 4 neutropenia lasting >7 days; (2) Febrile neutropenia, defined as absolute neutrophil count (ANC) <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than 1 hour; (3) Grade >=3 neutropenic infection; (4) Grade >=3 thrombocytopenia with bleeding; (5) Grade 4 thrombocytopenia. Non-Hematologic: (1) Grade >=3 non laboratory toxicities (excluding infusion reactions), except those that had not been maximally treated (eg, nausea, vomiting, diarrhea); (2) Grade >=3 laboratory abnormalities (other than aspartate aminotransferase [AST]/alanine aminotransferase [ALT]) if: Medical intervention was required to treat the participant, or The abnormality led to hospitalization; (3) Grade 4 AST and ALT increase.
Time Frame: First 2 Cycles (28 days in each cycle)
Population: All enrolled participants who were eligible for the study and received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities)
Description: An AE was any untoward medical occurrence in a participant administered a product or medical device without regard to possibility of causal relationship. Serious AEs (SAEs) were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions); resulted in congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. AEs were graded by the investigator according to NCI CTCAE version 4.03 (Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE). AEs included non-serious AEs and SAEs.
Time Frame: Day 1 up to 60 days after last dose of study treatment
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants
  AEs | 11 | 6 | 4 | 3
  SAEs | 3 | 3 | 2 | 2
  Grade 3 or 4 | 2 | 3 | 2 | 1
  Grade 5 | 0 | 2 | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (PF-05082566 Related)
Description: An AE was any untoward medical occurrence in a participant administered a product or medical device has a causal relationship with PF-05082566. SAEs were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions); resulted in congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. AEs were graded by the investigator according to NCI CTCAE version 4.03 (Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE). AEs included non-serious AEs and SAEs.
Time Frame: Day 1 up to 60 days after last dose of study treatment
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants
  AEs | 7 | 6 | 3 | 3
  SAEs | 0 | 0 | 0 | 0
  Grade 3 or 4 AEs | 0 | 2 | 0 | 0
  Grade 5 AEs | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Mogamulizumab Related)
Description: An AE was any untoward medical occurrence in a participant administered a product or medical device has a causal relationship with Mogamulizumab. SAEs were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions); resulted in congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. AEs were graded by the investigator according to NCI CTCAE version 4.03 (Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE). AEs included non-serious AEs and SAEs.
Time Frame: Day 1 up tp 60 days after last dose of study treatment
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants
  AEs | 7 | 6 | 4 | 3
  SAEs | 0 | 0 | 0 | 0
  Grade 3 or 4 AEs | 0 | 2 | 0 | 0
  Grade 5 AEs | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities as Characterized by Type, Frequency, Severity (as Graded by NCI CTCAE) -Grades 3 or 4
Description: The hematology laboratory tests include: Anemia, Hemoglobin increased, Lymphocyte count increased, Lymphopenia, Neutrophils (absolute), Platelets, White blood cells.
Time Frame: Screening (within 28 days prior to registration) up to 28 days (+7 days) after the last dose of study treatment
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants
  Anemia | 1 | 1 | 0 | 0
  Hemoglobin increased | 0 | 0 | 0 | 0
  Lymphocyte count increased | 0 | 0 | 0 | 0
  Lymphopenia | 6 | 0 | 2 | 0
  Neutrophils (absolute) | 0 | 0 | 0 | 0
  Platelets | 0 | 0 | 0 | 0
  White blood cells | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Chemistries Laboratory Abnormalities as Characterized by Type, Frequency, Severity (as Graded by NCI CTCAE) -Grades 3 or 4
Description: The chemistry laboratory tests included: Alanine aminotransferase, Aspartate Aminotransferase, Alkaline Phosphatase, Lactate Dehydrogenase, Sodium, Potassium, Magnesium, Total Calcium, Phosphorus or Phosphate, Total bilirubin, Creatinine or creatinine clearance, Albumin, Total proteins, Uric Acid, BUN or Urea, Immunoglobulin G, Glucose (fasted).
Time Frame: Screening (within 28 days prior to registration) up to 28 days (+7 days) after the last dose of study treatment
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants
  ALT | 0 | 0 | 0 | 0
  Alkaline phosphatase | 0 | 0 | 0 | 0
  AST | 0 | 0 | 0 | 0
  Bilirubin (total) | 0 | 0 | 0 | 0
  Creatinine | 0 | 0 | 0 | 0
  Hypercalcemia | 0 | 0 | 0 | 0
  Hyperglycemia | 1 | 1 | 1 | 0
  Hyperkalemia | 0 | 0 | 0 | 0
  Hypermagnesemia | 0 | 0 | 0 | 0
  Hypernatremia | 0 | 0 | 0 | 0
  Hypoalbuminemia | 0 | 0 | 0 | 0
  Hypocalcemia | 0 | 0 | 0 | 0
  Hypoglycemia | 0 | 0 | 0 | 0
  Hypokalemia | 0 | 0 | 0 | 0
  Hypomagnesemia | 0 | 0 | 0 | 0
  Hyponatremia | 1 | 0 | 0 | 0
  Hypophosphatemia | 1 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinical Significant Observations in Vital Signs
Description: Blood pressure (BP) and pulse rate were recorded in supine or sitting position.
Time Frame: Screening (within 28 days prior to registration) up to 28 days (+7 days) after the last dose of study treatment
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Significant Changes From Baseline in Physical Examination
Description: Physical examination included an examination of major body systems, including general, head, ears, eyes, nose, mouth, throat, neck, lungs, heart, abdomen, musculoskeletal, lymph nodes, neurological and external genitalia. Significant changes from baseline were reported in each category.
Time Frame: Cycle 2 Day 1; End of the treatment.
Population: All enrolled participants who received at least 1 dose of study treatment. Number analyzed was the number of participants at the given category.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants
  Cycle 2 Day 1: number analyzed (Participants) | 11 | 5 | 3 | 3
  Cycle 2 Day 1 | 1 | 1 | 1 | 0
  End of Treatment: number analyzed (Participants) | 10 | 4 | 2 | 3
  End of Treatment | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Shift to Grades 2, 3, 4 or 5
Description: ECOG performance status was classified as 5 grades: 0 (Fully active, able to carry on all predisease performance without restriction); 1 (Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, ie, light house work, office work); 2 (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours); 3 (Capable of only limited self care, confined to bed or chair more than 50% of waking hours); 4 (Completely disabled. Cannot carry on any self care. Totally confined to bed or chair); 5 (Death). On-study shifts to ECOG performance statuses of 2, 3, 4 or 5 were reported.
Time Frame: Screening (within 28 days prior to registration) up to 28 days (+7 days) after the last dose of study treatment
Population: All enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-05082566-Cycle 5
Description: Maximum Observed Serum Concentration (Cmax) was observed directly from the data.
Time Frame: Cycle 5: Day 1 at pre-dose, at the end of PF-05082566 infusion, and at 2, 6, 168 hours (Day 8) and 336 hours (Day 15) after the start of PF-05082566 infusion.
Population: The PK parameter analysis population was defined as all enrolled participants who had been treated and whose concentration time data allowed the estimation of at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2
μg/mL | 18.71 (NA) — fewer than 3 participants had reportable parameter values | 27.80 (NA) — fewer than 3 participants had reportable parameter values |  | 105.7 (NA) — fewer than 3 participants had reportable parameter values

11. Secondary Outcome: Dose Normalized Cmax of PF-05082566-Cycle 5
Description: Dose normalized Cmax was calculated by Cmax / Dose
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL/mg/kg
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2
µg/mL/mg/kg | 15.61 (NA) — fewer than 3 participants had reportable parameter values | 25.60 (NA) — fewer than 3 participants had reportable parameter values |  | 21.13 (NA) — fewer than 3 participants had reportable parameter values

12. Secondary Outcome: Cmax of Mogamulizumab-Cycles 1 and 5
Description: Maximum Observed Serum Concentration (Cmax) was observed directly from the data.
Time Frame: Cycle 1: pre-dose and at the end of mogamulizumab infusion on Days 1, 8, 15 and 22; Cycle 5: Pre-dose, at the end of mogamulizumab infusion, and at 6 hours, 168 hours (Day 8) after the start of the mogamulizumab infusion; Pre-dose on Day 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 5 | 4 | 3
μg/mL
  Cycle 1 | 18.78 (19) | 19.73 (32) | 19.77 (16) | 19.82 (19)
  Cycle 5: number analyzed (Participants) | 2 | 1 | 0 | 2
  Cycle 5 | 31.05 (NA) — fewer than 3 participants had reportable parameter values | 31.90 (NA) — fewer than 3 participants had reportable parameter values |  | 32.62 (NA) — fewer than 3 participants had reportable parameter values

13. Secondary Outcome: Pre-dose Concentration During Multiple Dosing (Ctrough) of PF-05082566-Cycle 5
Description: Pre-dose Concentration during Multiple Dosing (Ctrough) was observed directly from data
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 1 | 1 | 0 | 2
μg/mL | 1.300 (NA) — fewer than 3 participants had reportable parameter values | 1.160 (NA) — fewer than 3 participants had reportable parameter values |  | 3.464 (NA) — fewer than 3 participants had reportable parameter values

14. Secondary Outcome: Ctrough of Mogamulizumab- Cycle 5
Description: Pre-dose Concentration during Multiple Dosing (Ctrough) was observed directly from data.
Time Frame: Cycle 5: Pre-dose, at the end of mogamulizumab infusion, and at 6 hours, 168 hours (Day 8) after the start of the mogamulizumab infusion; Pre-dose on Day 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2
μg/mL | 15.45 (NA) — fewer than 3 participants had reportable parameter values | 9.040 (NA) — fewer than 3 participants had reportable parameter values |  | 15.99 (NA) — fewer than 3 participants had reportable parameter values

15. Secondary Outcome: Time for Cmax (Tmax) of PF-05082566-Cycle 5
Description: Time for Cmax (Tmax) was observed directly from the data.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2
hour | 2.02 [2.00 to 2.03] | 6.00 [6.00 to 6.00] |  | 1.08 [1.00 to 1.25]

16. Secondary Outcome: Time of Last Measurable Concentration (Tlast) of PF-05082566-Cycle 5
Description: Time of last measurable concentration was observed directly from data.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2
hour | 336 [335 to 336] | 309 [309 to 309] |  | 97.6 [25.1 to 170]

17. Secondary Outcome: Tmax of Mogamulizumab-Cycles 1 and 5
Description: Time for Cmax (Tmax) was observed directly from the data.
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 5 | 4 | 3
hour
  Cycle 1 | 1.28 [1.00 to 5.50] | 1.30 [1.10 to 2.25] | 1.24 [1.15 to 4.58] | 1.03 [0.917 to 1.18]
  Cycle 5: number analyzed (Participants) | 2 | 1 | 0 | 2
  Cycle 5 | 13.5 [4.52 to 22.4] | 1.05 [1.05 to 1.05] |  | 1.05 [1.02 to 1.07]

18. Secondary Outcome: Tlast of Mogamulizumab-Cycles 1 and 5
Description: Time of last measurable concentration was observed directly from the data.
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 5 | 4 | 3
hour
  Cycle 1 | 166 [164 to 285] | 166 [163 to 214] | 143 [22.4 to 194] | 166 [166 to 171]
  Cycle 5: number analyzed (Participants) | 2 | 1 | 0 | 2
  Cycle 5 | 335 [334 to 335] | 308 [308 to 308] |  | 107 [45.2 to 168]

19. Secondary Outcome: Area Under the Serum Concentration-time Profile From Time 0 to the Time of the Last Measurable Concentration (AUClast) of PF-05082566-Cycle 5
Description: AUClast was area under the serum concentration-time profile from time 0 to the time of the last measurable concentration (Clast), which was measured by Linear/Log trapezoidal method.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2
μg*hr/mL | 1143 (NA) — fewer than 3 participants had reportable parameter values | 2700 (NA) — fewer than 3 participants had reportable parameter values |  | 3875 (NA) — fewer than 3 participants had reportable parameter values

20. Secondary Outcome: Dose Normalized AUClast of PF-05082566-Cycle 5
Description: Dose normalized AUClast was calculated by AUClast / Dose
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL/mg/kg
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2
µg•hr/mL/mg/kg | 952.5 (NA) — fewer than 3 participants had reportable parameter values | 2490 (NA) — fewer than 3 participants had reportable parameter values |  | 773.0 (NA) — fewer than 3 participants had reportable parameter values

21. Secondary Outcome: AUClast of Mogamulizumab-Cycles 1 and 5
Description: as for outcome 19
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 5 | 4 | 3
μg*hr/mL
  Cycle 1 | 2001 (24) | 2182 (36) | 1382 (133) | 2126 (24)
  Cycle 5: number analyzed (Participants) | 2 | 1 | 0 | 2
  Cycle 5 | 6853 (NA) — fewer than 3 participants had reportable parameter values | 5870 (NA) — fewer than 3 participants had reportable parameter values |  | 2310 (NA) — fewer than 3 participants had reportable parameter values

22. Secondary Outcome: Area Under the Serum Concentration-time Profile From Time 0 to 168 Hours (AUC168) of Mogamulizumab-Cycle 1
Description: AUC168 was area under the serum concentration-time profile from time 0 to 168 hours post dose (Cycle 1 only where dosing was once a week), which was measured by Linear/Log trapezoidal method.
Time Frame: Cycle 1: pre-dose and at the end of mogamulizumab infusion on Days 1, 8, 15 and 22
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 5 | 3 | 3
μg*hr/mL | 1945 (25) | 2124 (33) | 2353 (14) | 2123 (24)

23. Secondary Outcome: Area Under the Serum Concentration-time Profile From Time 0 to Time Tau (AUCtau) of Mogamulizumab-Cycle 5
Description: AUCtau was area under the serum concentration-time profile from time 0 to time tau, the dosing interval, where tau=336 hours
Time Frame: as for outcome 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 1
μg*hr/mL | 6868 (NA) — fewer than 3 participants had reportable parameter values | 6160 (NA) — fewer than 3 participants had reportable parameter values |  | 6950 (NA) — fewer than 3 participants had reportable parameter values

24. Secondary Outcome: Clearance (CL) of Mogamulizumab-Cycle 5
Description: Clearance (CL) was measured by Dose / AUCtau
Time Frame: as for outcome 14
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 1
mL/hr/kg | 0.146 (NA) — fewer than 3 participants had reportable parameter values | 0.162 (NA) — fewer than 3 participants had reportable parameter values |  | 0.144 (NA) — fewer than 3 participants had reportable parameter values

25. Secondary Outcome: Anti-Drug Antibody (ADA) Titer for PF-05082566
Description: Serum samples were assayed for ADA using a validated analytical method.
Time Frame: Pre-dose on Day 1 of Cycles 1, 3, 5, 8, 12, 16, 20, 24 up to 24 months
Population: Number of participants analyzed was determined as participants with treatment-induced ADA.
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 7 | 3 | 1 | 2
Titer | 14.98 [12.31 to 16.31] | 10.80 [6.23 to 10.92] | 17.25 [NA to NA] — Only 1 participant was positive for ADA | 8.03 [6.23 to 9.82]

26. Secondary Outcome: Neutralizing Antibodies (NAb) Titers for PF-05082566
Description: ADA positive samples were further analyzed for NAb using a validated assay.
Time Frame: Pre-dose on Day 1 of Cycles 1, 3, 5, 8, 12, 16, 20, 24 up to 24 months
Population: Number of participants analyzed was determined as participants with treatment-induced NAb.
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 7 | 2 | 1 | 1
Titer | 1.80 [1.56 to 1.86] | 1.30 [1.30 to 1.30] | 2.64 [NA to NA] — Only 1 participant was positive for NAb | 1.30 [NA to NA] — Only 1 participant was positive for NAb

27. Secondary Outcome: Anti-Drug Antibody (ADA) Titers for Mogamulizumab
Description: Serum samples were assayed for ADA using a validated analytical method.
Time Frame: Pre-dose on Day 1 of Cycles 1, 3, 5, 8, 12, 16, 20, 24 up to 24 months
Population: Number of participants analyzed was determined as participants with treatment-induced ADA.
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 0 | 1 | 0 | 0
Titer |  | 1024 [NA to NA] — Only 1 participant was positive for ADA |  |

28. Secondary Outcome: Neutralizing Antibodies (NAb) Titers for Mogamulizumab
Description: ADA positive samples were further analyzed for NAb using a validated assay
Time Frame: Pre-dose on Day 1 of Cycles 1, 3, 5, 8, 12, 16, 20, 24 up to 24 months
Population: Number of participants analyzed was determined as participants with treatment-induced NAb.
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

29. Secondary Outcome: Number of Participants With Objective Response (OR) and Immune-related Objective Response (irOR)
Description: OR was defined as best overall response (BOR) of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. Immune-related OR (irOR) was defined as immune-related BOR (irBOR) of immune-related CR (irCR) and immune-related PR (irPR) according to immune-related RECIST. CR: Complete disappearance of all target lesions with the exception of nodal disease; PR: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: Every 8 weeks up to 24 months
Population: The full analysis set included all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
Number analyzed (Participants) | 11 | 6 | 4 | 3
Participants
  Objective Response | 0 | 1 | 0 | 0
  immune-related Objective Response | 0 | 1 | 0 | 0

30. Secondary Outcome: Time to Response (TTR) and Immue-related Time to Response (irTTR)-Dose Expansion Portion
Description: TTR was defined, for participants with an OR, as the time from the date of first dose of study treatment to the first documentation of OR (CR or PR), which was subsequently confirmed. irTTR was defined, for participants with an irOR, as the time from the first dose of study treatment to the first documentation of irOR (irCR or irPR) which was subsequently confirmed. CR: Complete disappearance of all target lesions with the exception of nodal disease; PR: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: Every 8 weeks up to 24 months
Population: No participants were enrolled in the dose-expansion portion.
Groups:
- Dose Expansion Cohort: Expansion cohorts of participants were to be enrolled to further study the safety, tolerability, PK/PD, and preliminary anti tumor activity for PF-05082566 in combination with mogamulizumab, as well as to study tumor associated biomarkers.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

31. Secondary Outcome: Duration of Response (DR) and Immune-related DR (irDR) -Dose Expansion Portion
Description: DR was defined, for participants with an OR, as the time from first documentation of OR (CR or PR) to the date of first documentation of objective progression disease (PD) or death due to any cause. irDR was defined, for participants with an irOR, as the time from the first documentation of irOR (irCR or irPR) to the date of first documentation of immune-related PD (irPD) (which was subsequently confirmed) or death due to any cause. CR: Complete disappearance of all target lesions with the exception of nodal disease; PR: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions; PD: 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: Every 8 weeks from the first occurrence of CR or PR, until disease progression or death up to 24 months
Population: No participants were enrolled in the dose-expansion portion.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

32. Secondary Outcome: Progression Free Survival (PFS) and Immune-related PFS (irPFS) - Dose Expansion Portion
Description: PFS was defined as the time from the date of first dose of study treatment to the date of the first documentation of PD or death due to any cause, whichever occurred first. irPFS was defined as the time from the first dose of study treatment to the date of first documentation of irPD (which was subsequently confirmed) or death due to any cause, whichever occurred first. PD:20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: Every 8 weeks up to 24 months
Population: No participants were enrolled in the dose-expansion portion.
Arm/Group | Dose Expansion Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 60 days after last dose of study treatment
Arm/Group | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 100 mg + Mogamulizumab 1 mg/kg | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/11 | 3/6 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/11 | 3/6 | 2/4 | 2/3
Other Adverse Events (participants affected / at risk) | 11/11 | 6/6 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg (N=11) | PF-05082566 100 mg + Mogamulizumab 1 mg/kg (N=6) | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg (N=4) | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05082566 1.2 mg/kg + Mogamulizumab 1 mg/kg (N=11) | PF-05082566 100 mg + Mogamulizumab 1 mg/kg (N=6) | PF-05082566 2.4 mg/kg + Mogamulizumab 1 mg/kg (N=4) | PF-05082566 5 mg/kg + Mogamulizumab 1 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 1 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 5 | 2 | 2
Malaise (General disorders) | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 0 | 1
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 3 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to marginal efficacy and change in sponsor prioritization. No participants were enrolled in the dose-expansion portion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02444793/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT02444793/SAP_001.pdf